CLINICAL TRIAL: NCT01094184
Title: Open-Label Study of Bevacizumab (Avastin®) and Taxane Monotherapy for the First-Line Treatment of Patients With Advanced Triple Negative Breast Cancer
Brief Title: A Study of Bevacizumab With Taxane Therapy in Participants With Triple Negative Breast Cancer
Acronym: BATMAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22780; 2009-014279-37
Record Dates: First submitted 2010-03-16; First posted 2010-03-26 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel; Docetaxel

ARMS (2):
- Bevacizumab 10 mg/kg Q2W (Experimental): Participants will receive bevacizumab at a dose of 10 milligrams per kilogram (mg/kg) every 2 weeks (Q2W) as intravenous infusion along with paclitaxel every week (Q1W) or docetaxel every 3 weeks (Q3W) as per discretion of the treating physician until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Docetaxel
- Bevacizumab 15 mg/kg Q3W (Experimental): Participants will receive bevacizumab at a dose of 15 mg/kg Q3W as intravenous infusion along with paclitaxel Q1W or docetaxel Q3W as per discretion of the treating physician until disease progression, unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Docetaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 10 mg/kg Q2W or 15 mg/kg Q3W as intravenous infusion.
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel will be administered as intravenous infusion Q1W as per discretion of the treating physician.
Drug: Docetaxel — Docetaxel will be administered as intravenous infusion Q3W as per discretion of the treating physician. Protocol amendment 2 (dated 17-Feb-2011) removed the option to choose docetaxel.

SUMMARY:
This open-label, multi-center study will evaluate the safety, tolerability and effect of bevacizumab (Avastin) in combination with taxane (paclitaxel/ docetaxel) monotherapy on disease progression, survival time and Karnofsky performance status in female participants with estrogen-, progesterone- and human epidermal growth factor receptor 2 (HER2)-negative (triple-negative) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed triple-negative (estrogen, progesterone, and HER-2 receptor negative) adenocarcinoma of the breast in pre- or post-menopausal women with measurable or non-measurable metastatic disease
* Participant who in the Investigator's opinion requires combination therapy for their disease
* Life expectancy of greater than or equal to (>/=)12 weeks

Exclusion Criteria:

* Previous chemotherapy for metastatic breast cancer
* Participants currently undergoing radiation therapy for the treatment of metastatic disease (apart from the relief of metastatic bone pain)
* Major surgery or significant traumatic injury within 28 days prior to enrollment or anticipation of the need for major surgery during study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United Kingdom (10):
  - Bangor
  - Cottingham
  - Exeter
  - Grimsby
  - Harrogate
  - Plymouth
  - Portsmouth
  - Preston
  - Somerset
  - Wolverhampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 53 participants were screened; 49 participants were eligible for the study and assigned to study treatment
Groups:
- Bevacizumab 10 mg/kg Q2W: Participants received bevacizumab at a dose of 10 milligrams per kilogram (mg/kg) every 2 weeks (Q2W) as intravenous infusion along with paclitaxel every week (Q1W) or docetaxel every 3 weeks (Q3W) as per discretion of the treating physician until disease progression, unacceptable toxicity or withdrawal of consent.
- Bevacizumab 15 mg/kg Q3W: Participants received bevacizumab at a dose of 15 mg/kg Q3W as intravenous infusion along with paclitaxel Q1W or docetaxel Q3W as per discretion of the treating physician until disease progression, unacceptable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Started | 36 | 13
Completed | 1 | 2
Not Completed | 35 | 11
Not completed — Death | 35 | 11

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least one dose of study medication (taxane [paclitaxel/ docetaxel] or bevacizumab).
Groups:
- Bevacizumab 10 mg/kg Q2W: Participants received bevacizumab at a dose of 10 mg/kg Q2W as intravenous infusion along with paclitaxel Q1W or docetaxel Q3W as per discretion of the treating physician until disease progression, unacceptable toxicity or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W | Total
Number analyzed (Participants) | 36 | 13 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (14.74) | 58.4 (9.22) | 54.2 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 13 | 49
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) Score at Cycle 2
Description: FACT-B is used for assessment of health-related quality of life (QoL) in participants with breast cancer. It consists of 36 items, summarized to 5 subscales: physical (7 items), functional (7 items), social/family (7 items); all 3 ranged from 0 to 28, emotional (6 items) ranging from 0 to 24, and breast cancer subscale (9 items) ranging from 0 to 36; high subscale score represents a better QoL. All single-item measures range from 0='Not at all' to 4='Very much'. Total possible score ranged from 0 to 144. High scale score represents a better QoL.
Time Frame: Baseline, Cycle 2 (Cycle length=2 and 3 weeks)
Population: Intent-to-treat (ITT) analysis population included all participants who received at least 1 dose of all study medication (taxane and bevacizumab). 'Overall Number of Participants Analyzed'=participants who completed the questionnaire at Baseline; 'Number Analyzed'=participants who completed the questionnaire at Baseline and at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 31 | 12
units on a scale
  Baseline | 98.3 (21.342) | 102.21 (21.036)
  Change at Cycle 2: number analyzed (Participants) | 25 | 6
  Change at Cycle 2 | 5.83 (17.027) | -2.48 (14.697)

2. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 3
Description: FACT-B is used for assessment of health-related QoL in participants with breast cancer. It consists of 36 items, summarized to 5 subscales: physical (7 items), functional (7 items), social/family (7 items); all 3 ranged from 0 to 28, emotional (6 items) ranging from 0 to 24, and breast cancer subscale (9 items) ranging from 0 to 36; high subscale score represents a better QoL. All single-item measures range from 0='Not at all' to 4='Very much'. Total possible score ranged from 0 to 144. High scale score represents a better QoL.
Time Frame: Baseline, Cycle 3 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 3
units on a scale |  | 14.56 (13.961)

3. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 4
Description: as for outcome 2
Time Frame: Baseline, Cycle 4 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 20 | 6
units on a scale | 1.29 (16.304) | 0.09 (12.275)

4. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 5
Description: as for outcome 2
Time Frame: Baseline, Cycle 5 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 5.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 2
units on a scale | -10.77 (11.677) | 4.50 (27.577)

5. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 6
Description: as for outcome 2
Time Frame: Baseline, Cycle 6 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 6 | 7
units on a scale | 9.47 (16.356) | 10.08 (21.868)

6. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 7
Description: as for outcome 2
Time Frame: Baseline, Cycle 7 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 7 | 1
units on a scale | -6.24 (13.220) | 1.83

7. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 8
Description: as for outcome 2
Time Frame: Baseline, Cycle 8 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 4
units on a scale | 15.01 (9.805) | 15.44 (19.979)

8. Primary Outcome: Change From Baseline in FACT-B Score At Cycle 9
Description: as for outcome 2
Time Frame: Baseline, Cycle 9 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 9.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 1
units on a scale | -2.43 (7.762) | 7.00

9. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 10
Description: as for outcome 2
Time Frame: Baseline, Cycle 10 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 10.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 5
units on a scale | 2.71 (20.075) | 4.61 (13.968)

10. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 11
Description: as for outcome 2
Time Frame: Baseline, Cycle 11 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 11.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 1
units on a scale | 6.67 (11.889) | 8.17

11. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 12
Description: as for outcome 2
Time Frame: Baseline, Cycle 12 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 1
units on a scale | 9.22 (8.720) | 21.89

12. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 13
Description: as for outcome 2
Time Frame: Baseline, Cycle 13 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 13.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 0
units on a scale | -8.00 (9.899) |

13. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 14
Description: as for outcome 2
Time Frame: Baseline, Cycle 14 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 14.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 1
units on a scale | 6.83 (5.897) | 2.33

14. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 15
Description: as for outcome 2
Time Frame: Baseline, Cycle 15 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 15.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 0
units on a scale | -6.67 (8.250) |

15. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 16
Description: as for outcome 2
Time Frame: Baseline, Cycle 16 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 16.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 0
units on a scale | 11.83 (12.790) |

16. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 17
Description: as for outcome 2
Time Frame: Baseline, Cycle 17 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 17.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 0
units on a scale | 22.63 (13.157) |

17. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 18
Description: as for outcome 2
Time Frame: Baseline, Cycle 18 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 18.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
units on a scale | 10.28 (19.878) | 5.33

18. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 20
Description: as for outcome 2
Time Frame: Baseline, Cycle 20 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 20.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 0
units on a scale | 20.06 (12.787) |

19. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 21
Description: as for outcome 2
Time Frame: Baseline, Cycle 21 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 21.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
units on a scale | 25.75 (5.303) | 10.33

20. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 22
Description: as for outcome 2
Time Frame: Baseline, Cycle 22 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 22.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | 13.67 |

21. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 23
Description: as for outcome 2
Time Frame: Baseline, Cycle 23 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 23.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
units on a scale | 9.67 (20.742) | 7.33

22. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 24
Description: as for outcome 2
Time Frame: Baseline, Cycle 24 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | 6.00 |

23. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 25
Description: as for outcome 2
Time Frame: Baseline, Cycle 25 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 25.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 11.33

24. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 26
Description: as for outcome 2
Time Frame: Baseline, Cycle 26 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 26.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | 3.22 |

25. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 27
Description: as for outcome 2
Time Frame: Baseline, Cycle 27 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 27.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 1
units on a scale | -26.78 | 12.33

26. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 28
Description: as for outcome 2
Time Frame: Baseline, Cycle 28 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 28.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 16.33

27. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 29
Description: as for outcome 2
Time Frame: Baseline, Cycle 29 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 29.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 1
units on a scale | -3.00 | 9.78

28. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 30
Description: as for outcome 2
Time Frame: Baseline, Cycle 30 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 30.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | -3.11 |

29. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 32
Description: as for outcome 2
Time Frame: Baseline, Cycle 32 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 32.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 10.33

30. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 36
Description: as for outcome 2
Time Frame: Baseline, Cycle 36 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 36.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 3.33

31. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 37
Description: as for outcome 2
Time Frame: Baseline, Cycle 37 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 37.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 5.33

32. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 39
Description: as for outcome 2
Time Frame: Baseline, Cycle 39 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 39.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 9.33

33. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 42
Description: as for outcome 2
Time Frame: Baseline, Cycle 42 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 42.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 10.33

34. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 44
Description: as for outcome 2
Time Frame: Baseline, Cycle 44 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 44.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 11.33

35. Primary Outcome: Change From Baseline in FACT-B Score at Cycle 46
Description: as for outcome 2
Time Frame: Baseline, Cycle 46 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 46.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 13.33

36. Primary Outcome: Change From Baseline in FACT-B Score at End of Study
Description: as for outcome 2
Time Frame: Baseline, end of study (4-6 weeks after the last bevacizumab infusion) (maximum up to 5 years and 9 months)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at End of Study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 14 | 7
units on a scale | -10.33 (13.509) | -1.01 (9.343)

37. Primary Outcome: Change From Baseline in Euro Quality of Life (EQ-5D) - Health State Questionnaire Score at Cycle 2
Description: EQ-5D: participant rated questionnaire to assess health-related QoL in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Cycle 2 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline and 'Number Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 31 | 10
units on a scale
  Baseline | 0.6391 (0.25595) | 0.8152 (0.12211)
  Change at Cycle 2: number analyzed (Participants) | 25 | 5
  Change at Cycle 2 | 0.1090 (0.23563) | -0.2074 (0.19784)

38. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 3
Description: as for outcome 37
Time Frame: Baseline, Cycle 3 (Cycle length=2 and 3 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | 0.1920

39. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 4
Description: as for outcome 37
Time Frame: Baseline, Cycle 4 (Cycle length=2 and 3 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 20 | 5
units on a scale | -0.0105 (0.28263) | -0.0906 (0.06661)

40. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 5
Description: as for outcome 37
Time Frame: Baseline, Cycle 5 (Cycle length=2 and 3 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 1
units on a scale | -0.1164 (0.10045) | 0.2280

41. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 6
Description: as for outcome 37
Time Frame: Baseline, Cycle 6 (Cycle length=2 and 3 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 6
units on a scale | 0.0474 (0.23827) | -0.0735 (0.24131)

42. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 7
Description: as for outcome 37
Time Frame: Baseline, Cycle 7 (Cycle length=2 and 3 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 7 | 0
units on a scale | -0.0331 (0.18865) |

43. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 8
Description: as for outcome 37
Time Frame: Baseline, Cycle 8 (Cycle length=2 and 3 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 6 | 3
units on a scale | 0.0627 (0.23917) | -0.0523 (0.05250)

44. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 9
Description: as for outcome 37
Time Frame: Baseline, Cycle 9 (Cycle length=2 and 3 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 0
units on a scale | -0.1904 (0.24194) |

45. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 10
Description: as for outcome 37
Time Frame: Baseline, Cycle 10 (Cycle length=2 and 3 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 3
units on a scale | 0.0253 (0.32169) | -0.0540 (0.24990)

46. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 11
Description: as for outcome 37
Time Frame: Baseline, Cycle 11 (Cycle length=2 and 3 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 0
units on a scale | 0.0018 (0.20907) |

47. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 12
Description: as for outcome 37
Time Frame: Baseline, Cycle 12 (Cycle length=2 and 3 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 1
units on a scale | 0.0997 (0.35679) | -0.0520

48. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 13
Description: as for outcome 37
Time Frame: Baseline, Cycle 13 (Cycle length=2 and 3 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 0
units on a scale | -0.0930 (0.13152) |

49. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 14
Description: as for outcome 37
Time Frame: Baseline, Cycle 14 (Cycle length=2 and 3 weeks)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 1
units on a scale | 0.0620 (0.11033) | -0.3320

50. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 15
Description: as for outcome 37
Time Frame: Baseline, Cycle 15 (Cycle length=2 and 3 weeks)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 0
units on a scale | 0.0175 (0.19021) |

51. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 16
Description: as for outcome 37
Time Frame: Baseline, Cycle 16 (Cycle length=2 and 3 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 0
units on a scale | 0.0060 (0.21806) |

52. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 17
Description: as for outcome 37
Time Frame: Baseline, Cycle 17 (Cycle length=2 and 3 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 0
units on a scale | 0.1057 (0.17756) |

53. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 18
Description: as for outcome 37
Time Frame: Baseline, Cycle 18 (Cycle length=2 and 3 weeks)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
units on a scale | 0.0970 (0.01414) | -0.1570

54. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 20
Description: as for outcome 37
Time Frame: Baseline, Cycle 20 (Cycle length=2 and 3 weeks)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 0
units on a scale | 0.1035 (0.19670) |

55. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 21
Description: as for outcome 37
Time Frame: Baseline, Cycle 21 (Cycle length=2 and 3 weeks)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
units on a scale | 0.2955 (0.26658) | -0.1570

56. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 22
Description: as for outcome 37
Time Frame: Baseline, Cycle 22 (Cycle length=2 and 3 weeks)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | 0.0710 |

57. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 23
Description: as for outcome 37
Time Frame: Baseline, Cycle 23 (Cycle length=2 and 3 weeks)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
units on a scale | 0.0625 (0.06293) | -0.2280

58. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 24
Description: as for outcome 37
Time Frame: Baseline, Cycle 24 (Cycle length=2 and 3 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | 0.0540 |

59. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 25
Description: as for outcome 37
Time Frame: Baseline, Cycle 25 (Cycle length=2 and 3 weeks)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.3320

60. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 26
Description: as for outcome 37
Time Frame: Baseline, Cycle 26 (Cycle length=2 and 3 weeks)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | 0.0180 |

61. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 27
Description: as for outcome 37
Time Frame: Baseline, Cycle 27 (Cycle length=2 and 3 weeks)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 1
units on a scale | 0.0540 | -0.3320

62. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 28
Description: as for outcome 37
Time Frame: Baseline, Cycle 28 (Cycle length=2 and 3 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.2610

63. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 29
Description: as for outcome 37
Time Frame: Baseline, Cycle 29 (Cycle length=2 and 3 weeks)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 1
units on a scale | -0.0860 | -0.2610

64. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 30
Description: as for outcome 37
Time Frame: Baseline, Cycle 30 (Cycle length=2 and 3 weeks)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
units on a scale | 0.0540 |

65. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 32
Description: as for outcome 37
Time Frame: Baseline, Cycle 32 (Cycle length=2 and 3 weeks)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.2610

66. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 36
Description: as for outcome 37
Time Frame: Baseline, Cycle 36 (Cycle length=2 and 3 weeks)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.2610

67. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 37
Description: as for outcome 37
Time Frame: Baseline, Cycle 37 (Cycle length=2 and 3 weeks)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.2610

68. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 39
Description: as for outcome 37
Time Frame: Baseline, Cycle 39 (Cycle length=2 and 3 weeks)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.2610

69. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 40
Description: as for outcome 37
Time Frame: Baseline, Cycle 40 (Cycle length=2 and 3 weeks)
Population: ITT analysis population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants who completed the questionnaire at Baseline as well as at Cycle 40.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.2610

70. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 42
Description: as for outcome 37
Time Frame: Baseline, Cycle 42 (Cycle length=2 and 3 weeks)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.2610

71. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 44
Description: as for outcome 37
Time Frame: Baseline, Cycle 44 (Cycle length=2 and 3 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.3320

72. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at Cycle 46
Description: as for outcome 37
Time Frame: Baseline, Cycle 46 (Cycle length=2 and 3 weeks)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
units on a scale |  | -0.3320

73. Primary Outcome: Change From Baseline in EQ-5D- Health State Questionnaire Score at End of Study
Description: as for outcome 37
Time Frame: Baseline, end of study (4-6 weeks after the last bevacizumab infusion) (maximum up to 5 years and 9 months)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 14 | 5
units on a scale | -0.1344 (0.20511) | -0.1178 (0.14225)

74. Primary Outcome: Change From Baseline in EQ-5D - Visual Analogue Scale (VAS) Score at Cycle 2
Description: EQ-5D: participant rated questionnaire to assess health-related QoL in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Cycle 2 (Cycle length=2 and 3 weeks)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 30 | 12
mm
  Baseline | 64.8 (24.34) | 60.3 (26.96)
  Change at Cycle 2: number analyzed (Participants) | 23 | 6
  Change at Cycle 2 | -1.0 (18.59) | -8.3 (19.41)

75. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 3
Description: as for outcome 74
Time Frame: Baseline, Cycle 3 (Cycle length=2 and 3 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 3
mm |  | 20.0 (26.46)

76. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 4
Description: as for outcome 74
Time Frame: Baseline, Cycle 4 (Cycle length=2 and 3 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 19 | 6
mm | -1.9 (18.23) | 3.3 (29.27)

77. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 5
Description: as for outcome 74
Time Frame: Baseline, Cycle 5 (Cycle length=2 and 3 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 2
mm | -8.2 (17.57) | 7.0 (46.67)

78. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 6
Description: as for outcome 74
Time Frame: Baseline, Cycle 6 (Cycle length=2 and 3 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 6 | 7
mm | 9.8 (22.00) | 21.4 (35.69)

79. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 7
Description: as for outcome 74
Time Frame: Baseline, Cycle 7 (Cycle length=2 and 3 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 1
mm | -3.6 (12.10) | -9.0

80. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 8
Description: as for outcome 74
Time Frame: Baseline, Cycle 8 (Cycle length=2 and 3 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 3
mm | 11.0 (27.60) | 35.0 (22.91)

81. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 9
Description: as for outcome 74
Time Frame: Baseline, Cycle 9 (Cycle length=2 and 3 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 2
mm | -5.8 (15.43) | 27.5 (45.96)

82. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 10
Description: as for outcome 74
Time Frame: Baseline, Cycle 10 (Cycle length=2 and 3 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 5
mm | 6.0 (21.91) | 14.0 (32.79)

83. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 11
Description: as for outcome 74
Time Frame: Baseline, Cycle 11 (Cycle length=2 and 3 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 5 | 1
mm | 2.0 (24.14) | 40.0

84. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 12
Description: as for outcome 74
Time Frame: Baseline, Cycle 12 (Cycle length=2 and 3 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 1
mm | 13.7 (24.19) | 60.0

85. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 13
Description: as for outcome 74
Time Frame: Baseline, Cycle 13 (Cycle length=2 and 3 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 0
mm | -3.0 (2.83) |

86. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 14
Description: as for outcome 74
Time Frame: Baseline, Cycle 14 (Cycle length=2 and 3 weeks)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 1
mm | -5.0 (20.00) | 9.0

87. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 15
Description: as for outcome 74
Time Frame: Baseline, Cycle 15 (Cycle length=2 and 3 weeks)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 0
mm | 5.0 (7.07) |

88. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 16
Description: as for outcome 74
Time Frame: Baseline, Cycle 16 (Cycle length=2 and 3 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 0
mm | 7.3 (37.87) |

89. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 17
Description: as for outcome 74
Time Frame: Baseline, Cycle 17 (Cycle length=2 and 3 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 3 | 0
mm | 30.0 (25.00) |

90. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 18
Description: as for outcome 74
Time Frame: Baseline, Cycle 18 (Cycle length=2 and 3 weeks)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
mm | 9.5 (55.86) | 10.0

91. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 20
Description: as for outcome 74
Time Frame: Baseline, Cycle 20 (Cycle length=2 and 3 weeks)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 4 | 0
mm | 15.0 (31.36) |

92. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 21
Description: as for outcome 74
Time Frame: Baseline, Cycle 21 (Cycle length=2 and 3 weeks)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
mm | 27.5 (31.82) | 8.0

93. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 22
Description: as for outcome 74
Time Frame: Baseline, Cycle 22 (Cycle length=2 and 3 weeks)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
mm | 52.0 |

94. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 23
Description: as for outcome 74
Time Frame: Baseline, Cycle 23 (Cycle length=2 and 3 weeks)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 2 | 1
mm | 23.5 (47.38) | 10.0

95. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 24
Description: as for outcome 74
Time Frame: Baseline, Cycle 24 (Cycle length=2 and 3 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
mm | -20.0 |

96. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 25
Description: as for outcome 74
Time Frame: Baseline, Cycle 25 (Cycle length=2 and 3 weeks)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 9.0

97. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 26
Description: as for outcome 74
Time Frame: Baseline, Cycle 26 (Cycle length=2 and 3 weeks)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
mm | -20.0 |

98. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 27
Description: as for outcome 74
Time Frame: Baseline, Cycle 27 (Cycle length=2 and 3 weeks)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 1
mm | -20.0 | 10.0

99. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 28
Description: as for outcome 74
Time Frame: Baseline, Cycle 28 (Cycle length=2 and 3 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 9.0

100. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 29
Description: as for outcome 74
Time Frame: Baseline, Cycle 29 (Cycle length=2 and 3 weeks)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 1
mm | -20.0 | 10.0

101. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 30
Description: as for outcome 74
Time Frame: Baseline, Cycle 30 (Cycle length=2 and 3 weeks)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 1 | 0
mm | -20.0 |

102. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 32
Description: as for outcome 74
Time Frame: Baseline, Cycle 32 (Cycle length=2 and 3 weeks)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 9.0

103. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 36
Description: as for outcome 74
Time Frame: Baseline, Cycle 36 (Cycle length=2 and 3 weeks)
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 8.0

104. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 37
Description: as for outcome 74
Time Frame: Baseline, Cycle 37 (Cycle length=2 and 3 weeks)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 8.0

105. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 39
Description: as for outcome 74
Time Frame: Baseline, Cycle 39 (Cycle length=2 and 3 weeks)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 8.0

106. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 40
Description: as for outcome 74
Time Frame: Baseline, Cycle 40 (Cycle length=2 and 3 weeks)
Population: as for outcome 69
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 5.0

107. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 42
Description: as for outcome 74
Time Frame: Baseline, Cycle 42 (Cycle length=2 and 3 weeks)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 7.0

108. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 44
Description: as for outcome 74
Time Frame: Baseline, Cycle 44 (Cycle length=2 and 3 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 13.0

109. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at Cycle 46
Description: as for outcome 74
Time Frame: Baseline, Cycle 46 (Cycle length=2 and 3 weeks)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 0 | 1
mm |  | 14.0

110. Primary Outcome: Change From Baseline in EQ-5D-VAS Score at End of Study
Description: as for outcome 74
Time Frame: Baseline, end of study (4-6 weeks after the last bevacizumab infusion) (maximum up to 5 years and 9 months)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 12 | 7
mm | -2.7 (13.17) | -1.4 (22.34)

111. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause
Time Frame: Baseline up to death (overall approximately 5 years and 9 months)
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 35 | 13
percentage of participants | 97.1 | 84.6

112. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from start of taxane plus bevacizumab therapy to death due to any cause. Overall survival was calculated in months as (date of death from any cause - date of first administration of taxane or bevacizumab + 1) / 30.4375 and rounded to 1 decimal place. Participants for whom no death was captured on the clinical database were censored at the last date they were known to be alive.
Time Frame: Baseline up to death (overall approximately 5 years and 9 months)
Population: ITT analysis population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 35 | 13
months | 11.6 [8.5 to 16.9] | 18.9 [12.8 to 33.6]

113. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Disease progression was defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 mm of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Time Frame: Baseline up to disease progression (overall approximately 5 years and 9 months)
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 35 | 13
percentage of participants | 74.3 | 69.2

114. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from the start of taxane plus bevacizumab therapy to investigator assessed disease progression and was calculated in months as (date of Investigator assessed disease progression - date of first administration of taxane or bevacizumab + 1) / 30.4375 and rounded to 1 decimal place. Participants who had not progressed at the time of study completion (including participants who had died before progressive disease) or who were lost to follow-up were censored at the last bevacizumab administration date. Disease progression was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Time Frame: Baseline up to disease progression (overall approximately 5 years and 9 months)
Population: ITT analysis population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 35 | 13
months | 6.7 [4.5 to 14.1] | 7.9 [3.2 to 9.7]

115. Secondary Outcome: Percentage of Participants By Karnofsky Performance Status Scale Scores
Description: Karnofsky performance score is used to quantify participant's general well-being and activities of daily life and participants are classified based on their functional impairment. Karnofsky performance score is 11 level score which range between 0% (death) to 100% (no evidence of disease). Higher score means higher ability to perform daily tasks.
Time Frame: Baseline, Cycle 1 thereafter every cycle up to Cycle 47 (Cycle length=2 and 3 weeks), end of study (4-6 weeks after the last bevacizumab infusion) (maximum up to 5 years and 9 months)
Population: ITT analysis population. Here, 'Number Analyzed' signifies the number of participants who underwent Karnofsky Performance Status Scale Score assessment at specified time points for different arms, respectively. Data is not reported for Cycles 35, 41, 44 as no participant was evaluable at these time points.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Number analyzed (Participants) | 35 | 13
percentage of participants
  Baseline, 60%: number analyzed (Participants) | 33 | 12
  Baseline, 60% | 3.0 | 8.0
  Baseline, 70%: number analyzed (Participants) | 33 | 12
  Baseline, 70% | 9.0 | 8.0
  Baseline, 80%: number analyzed (Participants) | 33 | 12
  Baseline, 80% | 27.0 | 25.0
  Baseline, 90%: number analyzed (Participants) | 33 | 12
  Baseline, 90% | 30.0 | 25.0
  Baseline, 100%: number analyzed (Participants) | 33 | 12
  Baseline, 100% | 30.0 | 33.0
  Cycle 1, 60%: number analyzed (Participants) | 31 | 12
  Cycle 1, 60% | 6.0 | 0.0
  Cycle 1, 70%: number analyzed (Participants) | 31 | 12
  Cycle 1, 70% | 6.0 | 25.0
  Cycle 1, 80%: number analyzed (Participants) | 31 | 12
  Cycle 1, 80% | 26.0 | 25.0
  Cycle 1, 90%: number analyzed (Participants) | 31 | 12
  Cycle 1, 90% | 32.0 | 25.0
  Cycle 1, 100%: number analyzed (Participants) | 31 | 12
  Cycle 1, 100% | 29.0 | 25.0
  Cycle 2, 60%: number analyzed (Participants) | 31 | 10
  Cycle 2, 60% | 0.0 | 10.0
  Cycle 2, 70%: number analyzed (Participants) | 31 | 10
  Cycle 2, 70% | 13.0 | 30.0
  Cycle 2, 80%: number analyzed (Participants) | 31 | 10
  Cycle 2, 80% | 23.0 | 20.0
  Cycle 2, 90%: number analyzed (Participants) | 31 | 10
  Cycle 2, 90% | 35.0 | 30.0
  Cycle 2, 100%: number analyzed (Participants) | 31 | 10
  Cycle 2, 100% | 29.0 | 10.0
  Cycle 3, 70%: number analyzed (Participants) | 28 | 10
  Cycle 3, 70% | 4.0 | 30.0
  Cycle 3, 80%: number analyzed (Participants) | 28 | 10
  Cycle 3, 80% | 43.0 | 30.0
  Cycle 3, 90%: number analyzed (Participants) | 28 | 10
  Cycle 3, 90% | 32.0 | 30.0
  Cycle 3, 100%: number analyzed (Participants) | 28 | 10
  Cycle 3, 100% | 21.0 | 10.0
  Cycle 4, 60%: number analyzed (Participants) | 24 | 8
  Cycle 4, 60% | 0.0 | 13.0
  Cycle 4, 70%: number analyzed (Participants) | 24 | 8
  Cycle 4, 70% | 8.0 | 13.0
  Cycle 4, 80%: number analyzed (Participants) | 24 | 8
  Cycle 4, 80% | 29.0 | 38.0
  Cycle 4, 90%: number analyzed (Participants) | 24 | 8
  Cycle 4, 90% | 42.0 | 25.0
  Cycle 4, 100%: number analyzed (Participants) | 24 | 8
  Cycle 4, 100% | 21.0 | 13.0
  Cycle 5, 60%: number analyzed (Participants) | 19 | 9
  Cycle 5, 60% | 0.0 | 11.0
  Cycle 5, 70%: number analyzed (Participants) | 19 | 9
  Cycle 5, 70% | 5.0 | 11.0
  Cycle 5, 80%: number analyzed (Participants) | 19 | 9
  Cycle 5, 80% | 37.0 | 33.0
  Cycle 5, 90%: number analyzed (Participants) | 19 | 9
  Cycle 5, 90% | 42.0 | 33.0
  Cycle 5, 100%: number analyzed (Participants) | 19 | 9
  Cycle 5, 100% | 16.0 | 11.0
  Cycle 6, 80%: number analyzed (Participants) | 15 | 8
  Cycle 6, 80% | 33.0 | 50.0
  Cycle 6, 90%: number analyzed (Participants) | 15 | 8
  Cycle 6, 90% | 47.0 | 38.0
  Cycle 6, 100%: number analyzed (Participants) | 15 | 8
  Cycle 6, 100% | 20.0 | 13.0
  Cycle 7, 80%: number analyzed (Participants) | 14 | 7
  Cycle 7, 80% | 14.0 | 43.0
  Cycle 7, 90%: number analyzed (Participants) | 14 | 7
  Cycle 7, 90% | 64.0 | 29.0
  Cycle 7, 100%: number analyzed (Participants) | 14 | 7
  Cycle 7, 100% | 21.0 | 29.0
  Cycle 8, 70%: number analyzed (Participants) | 10 | 7
  Cycle 8, 70% | 0.0 | 14.0
  Cycle 8, 80%: number analyzed (Participants) | 10 | 7
  Cycle 8, 80% | 20.0 | 29.0
  Cycle 8, 90%: number analyzed (Participants) | 10 | 7
  Cycle 8, 90% | 60.0 | 43.0
  Cycle 8, 100%: number analyzed (Participants) | 10 | 7
  Cycle 8, 100% | 20.0 | 14.0
  Cycle 9, 60%: number analyzed (Participants) | 10 | 6
  Cycle 9, 60% | 0.0 | 17.0
  Cycle 9, 70%: number analyzed (Participants) | 10 | 6
  Cycle 9, 70% | 10.0 | 0.0
  Cycle 9, 80%: number analyzed (Participants) | 10 | 6
  Cycle 9, 80% | 10.0 | 17.0
  Cycle 9, 90%: number analyzed (Participants) | 10 | 6
  Cycle 9, 90% | 60.0 | 50.0
  Cycle 9, 100%: number analyzed (Participants) | 10 | 6
  Cycle 9, 100% | 20.0 | 17.0
  Cycle 10, 70%: number analyzed (Participants) | 11 | 5
  Cycle 10, 70% | 0.0 | 20.0
  Cycle 10, 80%: number analyzed (Participants) | 11 | 5
  Cycle 10, 80% | 9.0 | 40.0
  Cycle 10, 90%: number analyzed (Participants) | 11 | 5
  Cycle 10, 90% | 73.0 | 20.0
  Cycle 10, 100%: number analyzed (Participants) | 11 | 5
  Cycle 10, 100% | 18.0 | 20.0
  Cycle 11, 70%: number analyzed (Participants) | 10 | 4
  Cycle 11, 70% | 0.0 | 25.0
  Cycle 11, 80%: number analyzed (Participants) | 10 | 4
  Cycle 11, 80% | 0.0 | 25.0
  Cycle 11, 90%: number analyzed (Participants) | 10 | 4
  Cycle 11, 90% | 80.0 | 25.0
  Cycle 11, 100%: number analyzed (Participants) | 10 | 4
  Cycle 11, 100% | 20.0 | 25.0
  Cycle 12, 70%: number analyzed (Participants) | 10 | 4
  Cycle 12, 70% | 0.0 | 25.0
  Cycle 12, 80%: number analyzed (Participants) | 10 | 4
  Cycle 12, 80% | 0.0 | 25.0
  Cycle 12, 90%: number analyzed (Participants) | 10 | 4
  Cycle 12, 90% | 80.0 | 25.0
  Cycle 12, 100%: number analyzed (Participants) | 10 | 4
  Cycle 12, 100% | 20.0 | 25.0
  Cycle 13, 90%: number analyzed (Participants) | 8 | 2
  Cycle 13, 90% | 88.0 | 100.0
  Cycle 13, 100%: number analyzed (Participants) | 8 | 2
  Cycle 13, 100% | 13.0 | 0.0
  Cycle 14, 80%: number analyzed (Participants) | 8 | 1
  Cycle 14, 80% | 13.0 | 0.0
  Cycle 14, 90%: number analyzed (Participants) | 8 | 1
  Cycle 14, 90% | 75.0 | 100.0
  Cycle 14, 100%: number analyzed (Participants) | 8 | 1
  Cycle 14, 100% | 13.0 | 0.0
  Cycle 15, 80%: number analyzed (Participants) | 7 | 1
  Cycle 15, 80% | 14.0 | 0.0
  Cycle 15, 90%: number analyzed (Participants) | 7 | 1
  Cycle 15, 90% | 71.0 | 100.0
  Cycle 15, 100%: number analyzed (Participants) | 7 | 1
  Cycle 15, 100% | 14.0 | 0.0
  Cycle 16, 80%: number analyzed (Participants) | 4 | 1
  Cycle 16, 80% | 25.0 | 0.0
  Cycle 16, 90%: number analyzed (Participants) | 4 | 1
  Cycle 16, 90% | 75.0 | 100.0
  Cycle 16, 100%: number analyzed (Participants) | 4 | 1
  Cycle 16, 100% | 0.0 | 0.0
  Cycle 17, 90%: number analyzed (Participants) | 4 | 1
  Cycle 17, 90% | 75.0 | 100.0
  Cycle 17, 100%: number analyzed (Participants) | 4 | 1
  Cycle 17, 100% | 25.0 | 0.0
  Cycle 18, 90%: number analyzed (Participants) | 4 | 1
  Cycle 18, 90% | 75.0 | 100.0
  Cycle 18, 100%: number analyzed (Participants) | 4 | 1
  Cycle 18, 100% | 25.0 | 0.0
  Cycle 19, 90%: number analyzed (Participants) | 4 | 1
  Cycle 19, 90% | 75.0 | 0.0
  Cycle 19, 100%: number analyzed (Participants) | 4 | 1
  Cycle 19, 100% | 25.0 | 100.0
  Cycle 20, 80%: number analyzed (Participants) | 4 | 1
  Cycle 20, 80% | 0.0 | 100.0
  Cycle 20, 90%: number analyzed (Participants) | 4 | 1
  Cycle 20, 90% | 75.0 | 0.0
  Cycle 20, 100%: number analyzed (Participants) | 4 | 1
  Cycle 20, 100% | 25.0 | 0.0
  Cycle 21, 90%: number analyzed (Participants) | 4 | 1
  Cycle 21, 90% | 50.0 | 100.0
  Cycle 21, 100%: number analyzed (Participants) | 4 | 1
  Cycle 21, 100% | 50.0 | 0.0
  Cycle 22, 90%: number analyzed (Participants) | 2 | 1
  Cycle 22, 90% | 50.0 | 100.0
  Cycle 22, 100%: number analyzed (Participants) | 2 | 1
  Cycle 22, 100% | 50.0 | 0.0
  Cycle 23, 90%: number analyzed (Participants) | 3 | 1
  Cycle 23, 90% | 67.0 | 100.0
  Cycle 23, 100%: number analyzed (Participants) | 3 | 1
  Cycle 23, 100% | 33.0 | 0.0
  Cycle 24, 90%: number analyzed (Participants) | 3 | 1
  Cycle 24, 90% | 67.0 | 100.0
  Cycle 24, 100%: number analyzed (Participants) | 3 | 1
  Cycle 24, 100% | 33.0 | 0.0
  Cycle 25, 90%: number analyzed (Participants) | 3 | 1
  Cycle 25, 90% | 67.0 | 100.0
  Cycle 25, 100%: number analyzed (Participants) | 3 | 1
  Cycle 25, 100% | 33.0 | 0.0
  Cycle 26, 90%: number analyzed (Participants) | 4 | 1
  Cycle 26, 90% | 75.0 | 100.0
  Cycle 26, 100%: number analyzed (Participants) | 4 | 1
  Cycle 26, 100% | 25.0 | 0.0
  Cycle 27, 90%: number analyzed (Participants) | 2 | 1
  Cycle 27, 90% | 50.0 | 100.0
  Cycle 27, 100%: number analyzed (Participants) | 2 | 1
  Cycle 27, 100% | 50.0 | 0.0
  Cycle 28, 90%: number analyzed (Participants) | 1 | 1
  Cycle 28, 90% | 100.0 | 100.0
  Cycle 28, 100%: number analyzed (Participants) | 1 | 1
  Cycle 28, 100% | 0.0 | 0.0
  Cycle 29, 90%: number analyzed (Participants) | 1 | 0
  Cycle 29, 90% | 100.0 |
  Cycle 30, 80%: number analyzed (Participants) | 1 | 0
  Cycle 30, 80% | 100.0 |
  Cycle 31, 90%: number analyzed (Participants) | 0 | 1
  Cycle 31, 90% |  | 100.0
  Cycle 32, 90%: number analyzed (Participants) | 0 | 1
  Cycle 32, 90% |  | 100.0
  Cycle 33, 90%: number analyzed (Participants) | 0 | 1
  Cycle 33, 90% |  | 100.0
  Cycle 34, 90%: number analyzed (Participants) | 0 | 1
  Cycle 34, 90% |  | 100.0
  Cycle 36, 90%: number analyzed (Participants) | 0 | 1
  Cycle 36, 90% |  | 100.0
  Cycle 37, 90%: number analyzed (Participants) | 0 | 1
  Cycle 37, 90% |  | 100.0
  Cycle 38, 90%: number analyzed (Participants) | 0 | 1
  Cycle 38, 90% |  | 100.0
  Cycle 39, 90%: number analyzed (Participants) | 0 | 1
  Cycle 39, 90% |  | 100.0
  Cycle 40, 90%: number analyzed (Participants) | 0 | 1
  Cycle 40, 90% |  | 100.0
  Cycle 42, 100%: number analyzed (Participants) | 0 | 1
  Cycle 42, 100% |  | 100.0
  Cycle 43, 100%: number analyzed (Participants) | 0 | 1
  Cycle 43, 100% |  | 100.0
  Cycle 45, 100%: number analyzed (Participants) | 0 | 1
  Cycle 45, 100% |  | 100.0
  Cycle 46, 100%: number analyzed (Participants) | 0 | 1
  Cycle 46, 100% |  | 100.0
  Cycle 47, 100%: number analyzed (Participants) | 0 | 1
  Cycle 47, 100% |  | 100.0
  End of Study, 50%: number analyzed (Participants) | 19 | 8
  End of Study, 50% | 5.0 | 0.0
  End of Study, 60%: number analyzed (Participants) | 19 | 8
  End of Study, 60% | 0.0 | 13.0
  End of Study, 70%: number analyzed (Participants) | 19 | 8
  End of Study, 70% | 16.0 | 25.0
  End of Study, 80%: number analyzed (Participants) | 19 | 8
  End of Study, 80% | 32.0 | 25.0
  End of Study, 90%: number analyzed (Participants) | 19 | 8
  End of Study, 90% | 42.0 | 38.0
  End of Study, 100%: number analyzed (Participants) | 19 | 8
  End of Study, 100% | 5.0 | 0.0

ADVERSE EVENTS:
Time Frame: Day 1 up to 6 months after last dose (overall approximately 5 years and 9 months)
Description: Treatment-emergent are events between first dose of study drug and up to 6 months after last dose that were absent before treatment or that worsened relative to pretreatment state. Safety analysis population.
Arm/Group | Bevacizumab 10 mg/kg Q2W | Bevacizumab 15 mg/kg Q3W
Serious Adverse Events (participants affected / at risk) | 15/36 | 7/13
Other Adverse Events (participants affected / at risk) | 35/36 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 10 mg/kg Q2W (N=36) | Bevacizumab 15 mg/kg Q3W (N=13)
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Catheter site dermatitis (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 10 mg/kg Q2W (N=36) | Bevacizumab 15 mg/kg Q3W (N=13)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 1
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 2 | 0
Hyphaema (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 3
Vision blurred (Eye disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 14 | 5
Diarrhoea (Gastrointestinal disorders) | 11 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 13 | 4
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 3
Toothache (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 1
Catheter site inflammation (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 26 | 9
Mucosal inflammation (General disorders) | 11 | 2
Oedema peripheral (General disorders) | 3 | 2
Pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 3 | 0
Ulcer (General disorders) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 3 | 0
Fungal infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 3
Nail infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2
Oral herpes (Infections and infestations) | 1 | 2
Paronychia (Infections and infestations) | 1 | 2
Tooth abscess (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 8 | 3
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 5 | 0
Weight increased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 3 | 0
White blood cells urine positive (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 11 | 3
Lethargy (Nervous system disorders) | 5 | 2
Neuralgia (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 17 | 8
Paraesthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 4 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 3 | 2
Breast pain (Reproductive system and breast disorders) | 2 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 3
Onycholysis (Skin and subcutaneous tissue disorders) | 6 | 2
Onychomadesis (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Flushing (Vascular disorders) | 2 | 0
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 9 | 4
Hypotension (Vascular disorders) | 2 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.